CLINICAL TRIAL: NCT00442624
Title: Effects of Chronic Insomnia on the Neuroendocrine Regulation of Glucose and Lipid Metabolism
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKBB 196/05 SB
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Insomnia
Keywords: insomnia; glucose metabolism; insulin resistance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with chronic insomnia
- 2: age, sex, bmi matched healthy controls

SUMMARY:
We aim to assess the influence of chronic insomnia on the neuroendocrine regulation of the glucose and lipid metabolism to more clearly define the metabolic derangements associated with chronic insomnia and to prove that chronic insomnia is associated with increased levels of stress hormones, cytokines and impaired insulin sensitivity.

DETAILED DESCRIPTION:
Sleep fragmentation has previously been shown to result in activation of the stress axis as indicated by enhanced cortisol and catecholamine release and a proinflammatory state mirrored by increased concentrations of proinflammatory cytokines such as IL-6 and TNFa. Therefore sleep deprivation is associated with a similar pattern of endocrine and proinflammatory alterations that may promote the insulin resistant state. Thus, it is of paramount interest to clearly define the metabolic alterations in patients with primary insomnia.

Patients with with suspected primary insomnia will be recruited from the sleep clinic at the University Hospital Basel and by newspaper ads. Primary insomnia will be diagnosed by a polysomnographic study and the exclusion of secondary causes such as depression, sleep apnea and restless legs syndrome. Eligible patients will be admitted to the CRC for metabolic studies, including baseline blood samples for the measurement of hormones, cytokines and adipokines, a euglycemic-hyperinsulinemic clamp study for the assessment of glucose turnover and insulin sensitivity and in vivo NMR studies to determine intrahepatic and intramyocellular lipid content.

The data obtained in insomnic patients will be compared to those of a control group matched for age, sex, BMI, menopausal status and physical activity selected from the general population.

ELIGIBILITY:
Inclusion Criteria:

• Patients with primary chronic insomnia based on clinical history and a polysomnographic study.

Exclusion Criteria:

* Diabetes mellitus
* Known other sleep disorders, such as depression, obstructive sleep apnea and restless legs syndrome
* Alcohol consumption > 40 g / d in males, > 20 g / d in females, respectively,
* Patients treated with medications potentially interfering with glucose metabolism, such as systemic steroids, immunosuppressive drugs (cyclosporine, tacrolimus, sirolimus), highly active antiretroviral therapy, hydrochlorothiazide > 25 mg/d
* Patients treated with lipid lowering drugs such as statins, fibrates, nicotinic acid derivatives, resins and ezetimibe in whom the lipid lowering therapy cannot be safely withheld for the duration of the study.
* Patients with LDL-cholesterol concentrations > 4.9 mmol/l and fasting triglyceride concentrations > 12 mmol/l.
* Any significant or unstable hepatic, cardiac, pulmonary, renal, neurological, musculoskeletal, hematological or endocrine disease.
* Pregnant or Breast Feeding women
* Woman of childbearing potential not using a reliable method of birth control such as oral contraceptives or IUD.
* History of claustrophobia
* Ferromagnetic implants including pacemakers.
* Subjects refusing or unable to give written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient clinic, general population
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-01; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bilz, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland